27/07/2023, V5

Cognitive Multisensory Rehabilitation for CRPS treatment

REC Ethics approval: 23/WS/0022 IRAS Project ID: 323695

Combe Park Bath BA3NG Telephone: 01225428331



## PARTICIPANT CONSENT FORM A: CRPS PATIENT

## COGNITIVE MULTISENSORY REHABILITATION, A NOVEL SENSORIMOTOR INTERVENTION FOR PAIN REDUCTION IN COMPLEX REGIONAL PAIN SYNDROME: A FEASIBILITY STUDY

Please initial either the YES or NO box

| | Name of researcher: Marc Aureli Pique Batalla | | |
|---|---|---|---|
| 1. | I confirm that I have read and understood the information sheet dated [20/07/2023, V5] for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. There will be 3 copies of this document: x1 copy for participant, x1 copy for medical records and x1 copy for investigator's site file. | YES | NO |
| 2. | I understand my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without my medical care and legal rights being affected. I understand that data collected prior to my withdrawal will be used in the study. | YES | NO |
| 3. | I understand that researchers from the Royal United Hospital (RUH; Marc Aureli Pique Batalla and Jenny Lewis), University of the West of England (UWE; Jenny Lewis), University of Bath (UoB; Janet Bultitude) and Cognitive Multisensory Rehabilitation Centre (Marco Rigoni) that are part of this study may examine and analyse data collected during the study. I give permission for these individuals to have access to this anonymised data. | YES | NO |
| 4. | I understand that all information and data collected from me, as part of the project will be securely retained by RUH for 5 years in line with NHS National record management guidelines. | YES YES | NO<br>NO |
| 5. | I consent to be audio recorded. | | |
| 6. | I confirm that my data, which will be anonymized, can be used for future undescribed analyses by researchers who may, but are not necessarily members of the named team of researchers responsible for the current study | YES | NO |
| 7. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from University of the West of England (UWE; Jenny Lewis), University of Bath (UoB; Janet Bultitude) and Cognitive Multisensory Rehabilitation Centre (Marco Rigoni), from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records | YES<br>YES | NO<br>NO |
| 8. | I agree to take part in the above study. | | |

27/07/2023, V5

Cognitive Multisensory Rehabilitation for CRPS treatment

REC Ethics approval: 23/WS/0022 IRAS Project ID: 323695

Combe Park Bath BA3NG Telephone: 01225428331



## Data protection

The Royal United Hospital (RUH) will process your data in accordance with the General Data Protection Regulation as applied, enacted and amended in UK law. Your data will only be processed with your consent for the purposes described above and will only be shared outside of Royal United Hospital (including overseas with appropriate safeguards) in the circumstances described above.

## Your rights

In respect of your personal data held by us, you have the following qualified rights to:

- access it
- receive it in a structured machine readable format
- rectify it if it is not accurate or complete
- erase it
- restrict its processing
- withdraw any consent provided or otherwise object to its processing
- complain to the Information Commissioner's Office (ICO)

To find out more or to exercise any of these rights please contact the Data Protection Officer via e-mail: <a href="mailto:dpo@ico.org.uk">dpo@ico.org.uk</a>

| Name of patient | Date | Signature |
|---|---|---|
| Name of person taking consent (If different from researcher) | Date | Signature |
| Name of researcher | Date | Signature |